CLINICAL TRIAL: NCT01093326
Title: Multicenter, Randomized, Double-blind, Parallel-group Extension to Study AC-058B201 to Investigate the Long-term Safety, Tolerability, and Efficacy of Three Doses of Ponesimod, an Oral S1P1 Receptor Agonist, in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Clinical Study to Investigate the Long-term Safety, Tolerability, and Efficacy of Ponesimod in Patients With Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-058B202; 2009-011470-15 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ponesimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ponesimod 10 mg (Experimental): Ponesimod 10 mg oral use
  Interventions: Drug: Ponesimod 10 mg
- Ponesimod 20 mg (Experimental): Ponesimod 20 mg oral use
  Interventions: Drug: Ponesimod 20 mg
- Ponesimod 40 mg (Experimental): Ponesimod 40 mg oral use
  Interventions: Drug: Ponesimod 40 mg

INTERVENTIONS:
Drug: Ponesimod 10 mg — Ponesimod 10 mg oral use
  Arms: Ponesimod 10 mg
Drug: Ponesimod 20 mg — Ponesimod 20 mg oral use
  Arms: Ponesimod 20 mg
Drug: Ponesimod 40 mg — Ponesimod 40 mg oral use
  Arms: Ponesimod 40 mg

SUMMARY:
This study is an extension to the study AC-058B201 and will investigate the long-term safety, tolerability and efficacy of ponesimod in patients with relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed study treatment at their regular Week 24 (End of treatment) visit within the core study AC-058B201.
2. Signed informed consent for participating in the extension study.

Exclusion Criteria:

1. Any clinically relevant medical or surgical condition, which, in the opinion of the investigator, would put the patient at risk by participating in the extension study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 353 (Actual)
Dates: Start 2010-05-12 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (16):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Palo Alto, California
  - Sacramento, California
  - Venice, Florida
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Lenexa, Kansas
  - Latham, New York
  - Schenectady, New York
  - Stony Brook, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Burlington, Vermont
  - Kirkland, Washington
- Vienna, Austria
- Sofia, Bulgaria
- Ottawa, Ontario, Canada
- Czechia (6):
  - Brno
  - Jihlava
  - Olomouc
  - Ostrava-Poruba
  - Prague
  - Teplice
- Finland (4):
  - Helsinki
  - Hyvinkää
  - Tampere
  - Turku
- Montpellier, France
- Germany (3):
  - Berlin
  - Essen
  - Ulm
- Hungary (4):
  - Budapest
  - Esztergom
  - Győr
  - Miskolc
- Israel (2):
  - Tel Litwinsky
  - Ẕerifin
- Breda, Netherlands
- Poland (4):
  - Katowice
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (2):
  - Cluj-Napoca
  - Timișoara
- Russia (8):
  - Kazan'
  - Moscow
  - Nizhny Novgorod
  - Pyatigorsk
  - Saint Petersburg
  - Samara
  - Saratov
  - Ufa
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Niš
- Spain (3):
  - Majadahonda
  - Málaga
  - Seville
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Umeå
- Lugano, Switzerland
- Ukraine (4):
  - Chernihiv
  - Dnipropetrovsk
  - Kyiv
  - Odesa
- United Kingdom (3):
  - Bristol
  - London
  - Plymouth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were enrolled in the core study (NCT01006265) entered this extension study. As planned, combined analysis (core plus extension study) was done for efficacy and safety (435 participants).
Pre-assignment Details: Data reported in each arm are based on first dose received during treatment period (TP) 1.
Groups:
- Ponesimod 10 Milligrams (mg): Participants with relapsing-remitting multiple sclerosis having completed their regular Week 24 treatment visit of the core study (NCT01006265) while receiving ponesimod 10 mg or placebo, entered this extension study and received ponesimod 10 mg capsules orally once daily during treatment period (TP) 1. Participants continued to receive ponesimod 10 mg tablet orally, once daily during TP2. All participants received ponesimod 20 mg tablet orally, once daily during TP3.
- Ponesimod 20 Milligrams (mg): Participants with relapsing-remitting multiple sclerosis having completed their regular Week 24 treatment visit of the core study (NCT01006265) while receiving ponesimod 20 mg or placebo, entered this extension study and received ponesimod 20 mg capsules orally once daily during TP1. Participants continued to receive ponesimod 20 mg tablet orally, once daily during TP2 and TP3.
- Ponesimod 40 Milligrams (mg): Participants with relapsing-remitting multiple sclerosis having completed their regular Week 24 treatment visit of the core study (NCT01006265) while receiving ponesimod 40 mg or placebo, entered this extension study and received ponesimod 40 mg capsules orally once daily during TP1. Participants were then re-randomized to receive ponesimod 10 or 20 mg tablet orally, once daily during TP2. All participants received ponesimod 20 mg tablet orally, once daily during TP3.
Period: Overall Study
Arm/Group | Ponesimod 10 Milligrams (mg) | Ponesimod 20 Milligrams (mg) | Ponesimod 40 Milligrams (mg)
Started | 115 | 121 | 117
Completed | 71 | 80 | 76
Not Completed | 44 | 41 | 41
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 7 | 6 | 3
Not completed — Lost to Follow-up | 2 | 5 | 4
Not completed — Physician Decision | 3 | 1 | 3
Not completed — Withdrawal by Subject | 30 | 27 | 26
Not completed — Adverse Event | 2 | 1 | 4
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponesimod 10 Milligrams (mg) | Ponesimod 20 Milligrams (mg) | Ponesimod 40 Milligrams (mg) | Total
Number analyzed (Participants) | 115 | 121 | 117 | 353
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 115 | 121 | 117 | 353
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (8.67) | 36.1 (8.58) | 35.9 (8.61) | 36.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 80 | 76 | 233
  Male | 38 | 41 | 41 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 115 | 121 | 115 | 351
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 9
  White | 112 | 118 | 110 | 340
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 4 | 2 | 2 | 8
  Bulgaria | 5 | 3 | 5 | 13
  Canada | 2 | 2 | 2 | 6
  Czech Republic | 12 | 17 | 14 | 43
  Finland | 6 | 6 | 4 | 16
  France | 1 | 1 | 1 | 3
  Germany | 1 | 1 | 2 | 4
  Hungary | 2 | 8 | 5 | 15
  Israel | 0 | 2 | 1 | 3
  Italy | 8 | 8 | 6 | 22
  Netherlands | 0 | 1 | 1 | 2
  Poland | 14 | 6 | 11 | 31
  Romania | 1 | 2 | 0 | 3
  Russia | 8 | 11 | 11 | 30
  Serbia | 16 | 13 | 11 | 40
  Spain | 1 | 4 | 4 | 9
  Sweden | 4 | 6 | 8 | 18
  Switzerland | 2 | 1 | 0 | 3
  Ukraine | 4 | 7 | 5 | 16
  United Kingdom | 5 | 4 | 5 | 14
  United States | 19 | 16 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) of Confirmed Relapses
Description: ARR is defined as the number of confirmed relapses per year. A relapse is defined as the occurrence of an acute episode of one or more new symptoms, or worsening of existing symptoms of multiple sclerosis (MS), not associated with fever or infection, and lasting for at least 24 hours after a stable period of at least 30 days. A confirmed relapse is a relapse accompanied by an increase from the previous clinically stable assessment (that is, performed at least 30 days after the onset of any previous relapse) of at least 0.5 point in the Expanded Disability Status Scale (EDSS) score, or one point in the score for at least one of the Functional System (FS) scores, excluding the bowel and bladder, and mental FS. EDSS is ordinal clinical scale ranges 0 (normal neurological examination) to 10 (death due to MS).
Time Frame: From ponesimod start date up to the end of Analysis Period (AP) 3. The actual time varied for each participant and could be up to 13.3 years
Population: Ponesimod analysis set (PAS) included all participants who received at least one dose of ponesimod at any time during the core and/or the extension study (435 participants).
Measure: Mean (95% Confidence Interval); unit: Confirmed relapses per year
Arm/Group | Ponesimod 10 Milligrams (mg) | Ponesimod 20 Milligrams (mg) | Ponesimod 40 Milligrams (mg)
Number analyzed (Participants) | 139 | 145 | 151
Confirmed relapses per year | 0.205 [0.150 to 0.282] | 0.142 [0.102 to 0.198] | 0.150 [0.105 to 0.215]

2. Primary Outcome: Time to First Confirmed Relapse
Description: Time to first confirmed relapse was reported. A relapse is defined as the occurrence of an acute episode of one or more new symptoms, or worsening of existing symptoms of multiple sclerosis (MS), not associated with fever or infection, and lasting for at least 24 hours after a stable period of at least 30 days. A confirmed relapse is a relapse accompanied by an increase from the previous clinically stable assessment (that is, performed at least 30 days after the onset of any previous relapse) of at least 0.5 point in the Expanded Disability Status Scale (EDSS) score, or one point in the score for at least one of the Functional System (FS) scores, excluding the bowel and bladder, and mental FS. EDSS is ordinal clinical scale ranges from 0 (normal neurological examination) to 10 (death due to MS).
Time Frame: as for outcome 1
Population: PAS included all participants who received at least one dose of ponesimod at any time during the core and/or the extension study (435 participants).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ponesimod 10 Milligrams (mg) | Ponesimod 20 Milligrams (mg) | Ponesimod 40 Milligrams (mg)
Number analyzed (Participants) | 139 | 145 | 151
Weeks | 272.3 [164.6 to NA] — NA indicates data for upper limit of 95% CI was not estimable due to less number of participants with event. | 656.7 [278.0 to NA] — NA indicates data for upper limit of 95% CI was not estimable due to less number of participants with event. | 431.7 [296.3 to NA] — NA indicates data for lower upper of 95% CI was not estimable due to less number of participants with event.

3. Primary Outcome: Time to 24 Weeks Confirmed Disability Progression
Description: Time to 24 weeks confirmed disability progression (accumulation) was reported. Disability progression is defined as an increase of at least 1 point in the EDSS score if baseline EDSS was between 1 and 5.0, an increase of at least 1.5 points if baseline EDSS was 0, or an increase of at least 0.5 points if the baseline EDSS was equal or greater than 5.5. A 24-week confirmed disability progression is defined as a 24-week sustained increase from baseline in the EDSS scores, that is, every EDSS score (scheduled or unscheduled, with or without relapse) within a 24-week duration after the first progression should meet the progression criteria as specified above. EDSS is ordinal clinical scale ranges from 0 (normal neurological examination) to 10 (death due to MS).
Time Frame: From ponesimod baseline up to the end of Analysis Period (AP) 3. The actual time varied for each participant and could be up to 13.3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ponesimod 10 Milligrams (mg) | Ponesimod 20 Milligrams (mg) | Ponesimod 40 Milligrams (mg)
Number analyzed (Participants) | 139 | 145 | 151
Weeks | NA [470.3 to NA] — NA indicates data for median and upper limit of 95% CI was not estimable due to less number of participants with event. | NA [NA to NA] — NA indicates data for median, upper, and lower limit of 95% CI was not estimable due to less number of participants with event. | NA [NA to NA] — NA indicates data for median, upper, and lower limit of 95% CI was not estimable due to less number of participants with event.

4. Other Pre Specified Outcome: Number of Participants With at Least One Treatment-emergent Serious Adverse Events (SAEs)
Description: Number of participants with at least one treatment-emergent SAEs were reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalisation; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important. Treatment-emergent SAEs were those SAEs that occurred at or after the initial administration of ponesimod up to 15 days (inclusive) after last administration of ponesimod as study drug.
Time Frame: From ponesimod start date up to the end of study treatment + 15 Days. The actual time of observation varied for each participant and could be up to 12.97 years + 15 days
Population: Ponesimod analysis set included all participants who received at least one dose of ponesimod at any time during the core and/or the extension study (435 participants).
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 10 Milligrams (mg) | Ponesimod 20 Milligrams (mg) | Ponesimod 40 Milligrams (mg)
Number analyzed (Participants) | 139 | 145 | 151
Participants | 32 | 35 | 25

ADVERSE EVENTS:
Time Frame: For Serious and Non-serious AEs: From ponesimod start date up to end of treatment + 15 days (up to 12.97 years + 15 days); For All-cause Mortality: From ponesimod start date to end of Analysis Period 3 (up to 13.3 years)
Description: Ponesimod analysis set included all participants who received at least one dose of ponesimod at any time during the core and/or the extension study (435 participants).
Arm/Group | Ponesimod 10 Milligrams (mg) | Ponesimod 20 Milligrams (mg) | Ponesimod 40 Milligrams (mg)
All-Cause Mortality (participants affected / at risk) | 0/139 | 1/145 | 0/151
Serious Adverse Events (participants affected / at risk) | 32/139 | 35/145 | 25/151
Other Adverse Events (participants affected / at risk) | 121/139 | 125/145 | 140/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponesimod 10 Milligrams (mg) (N=139) | Ponesimod 20 Milligrams (mg) (N=145) | Ponesimod 40 Milligrams (mg) (N=151)
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular Block Second Degree (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral Valve Prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract Nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular Hole (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular Oedema (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Maculopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Retinal Detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Rhegmatogenous Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Complicated Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Bone Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chemical Burn of Skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chest Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fracture Displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Magnetic Resonance Imaging Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of the Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Benign Hydatidiform Mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal Papilloma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0)
Altered State of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Postictal State (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tension Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Stress Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Intermenstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion Induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Oophorectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Varicose Vein (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponesimod 10 Milligrams (mg) (N=139) | Ponesimod 20 Milligrams (mg) (N=145) | Ponesimod 40 Milligrams (mg) (N=151)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 10 (15) | 7 (7)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 6 (9) | 8 (13)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 7 (18) | 8 (9)
Eye Pain (Eye disorders) | 7 (20) | 3 (4) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (8) | 4 (4) | 9 (9)
Constipation (Gastrointestinal disorders) | 4 (4) | 8 (8) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 12 (22) | 11 (13) | 9 (10)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (8) | 10 (10)
Toothache (Gastrointestinal disorders) | 6 (6) | 8 (9) | 9 (10)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4) | 4 (5)
Fatigue (General disorders) | 13 (15) | 18 (21) | 14 (21)
Oedema Peripheral (General disorders) | 3 (3) | 8 (8) | 16 (17)
Pyrexia (General disorders) | 5 (6) | 8 (8) | 7 (11)
Bronchitis (Infections and infestations) | 22 (38) | 22 (30) | 21 (30)
Conjunctivitis (Infections and infestations) | 9 (11) | 3 (5) | 2 (2)
Covid-19 (Infections and infestations) | 12 (13) | 19 (23) | 19 (23)
Cystitis (Infections and infestations) | 7 (14) | 8 (8) | 9 (15)
Gastroenteritis (Infections and infestations) | 11 (18) | 10 (15) | 7 (12)
Gastroenteritis Viral (Infections and infestations) | 5 (5) | 8 (14) | 5 (8)
Herpes Zoster (Infections and infestations) | 4 (4) | 9 (9) | 6 (6)
Influenza (Infections and infestations) | 20 (48) | 18 (51) | 20 (43)
Nasopharyngitis (Infections and infestations) | 46 (142) | 46 (106) | 45 (136)
Oral Herpes (Infections and infestations) | 9 (42) | 6 (12) | 9 (16)
Pharyngitis (Infections and infestations) | 12 (21) | 4 (4) | 7 (11)
Respiratory Tract Infection (Infections and infestations) | 12 (22) | 12 (13) | 9 (11)
Rhinitis (Infections and infestations) | 14 (21) | 12 (12) | 2 (2)
Sinusitis (Infections and infestations) | 12 (17) | 12 (26) | 15 (22)
Tonsillitis (Infections and infestations) | 7 (12) | 6 (7) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 27 (84) | 28 (87) | 39 (109)
Urinary Tract Infection (Infections and infestations) | 21 (79) | 21 (68) | 22 (45)
Viral Infection (Infections and infestations) | 7 (8) | 9 (19) | 8 (15)
Contusion (Injury, poisoning and procedural complications) | 9 (11) | 8 (12) | 8 (9)
Ligament Sprain (Injury, poisoning and procedural complications) | 7 (8) | 10 (12) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 16 (25) | 19 (38) | 19 (43)
Aspartate Aminotransferase Increased (Investigations) | 6 (7) | 10 (13) | 8 (17)
Blood Cholesterol Increased (Investigations) | 7 (14) | 4 (4) | 6 (9)
Forced Expiratory Volume Decreased (Investigations) | 14 (22) | 12 (23) | 17 (31)
Forced Vital Capacity Decreased (Investigations) | 9 (18) | 3 (4) | 7 (11)
Pulmonary Function Test Decreased (Investigations) | 5 (8) | 2 (3) | 8 (9)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 (16) | 16 (16) | 10 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 8 (8) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (28) | 16 (23) | 16 (22)
Back Pain (Musculoskeletal and connective tissue disorders) | 21 (26) | 23 (29) | 22 (31)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 (11) | 4 (4) | 8 (11)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 14 (16) | 9 (9)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 8 (10) | 8 (8)
Dizziness (Nervous system disorders) | 18 (18) | 14 (16) | 18 (24)
Headache (Nervous system disorders) | 38 (62) | 31 (79) | 41 (91)
Migraine (Nervous system disorders) | 9 (15) | 9 (13) | 12 (18)
Multiple Sclerosis (Nervous system disorders) | 7 (9) | 5 (5) | 1 (1)
Paraesthesia (Nervous system disorders) | 7 (12) | 7 (8) | 6 (8)
Anxiety (Psychiatric disorders) | 8 (12) | 9 (9) | 8 (10)
Depression (Psychiatric disorders) | 8 (8) | 11 (12) | 9 (13)
Insomnia (Psychiatric disorders) | 9 (10) | 11 (15) | 11 (14)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (18) | 13 (16) | 28 (37)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (14) | 21 (25)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (11) | 8 (9)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (13) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 9 (9) | 5 (6)
Hypertension (Vascular disorders) | 22 (24) | 19 (22) | 18 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT01093326/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT01093326/SAP_001.pdf